CLINICAL TRIAL: NCT03316534
Title: Effect of Aspirin on Abacavir-induced Platelet Reactivity in HIV-infected Patients
Acronym: ABC-ASA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera di Perugia (Other)
Responsible Party: Principal Investigator, Paolo Gresele, Full Professor, Internal Medicine, Azienda Ospedaliera di Perugia
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: 1452/13/ACC
Record Dates: First submitted 2017-10-12; First posted 2017-10-20 (Actual); Last update posted 2017-10-20 (Actual); Status verified 2017-10

CONDITIONS: HIV-infected Patients
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: HIV subjects (all on ABC therapy) who fulfilled thee admission criteria will be randomized to either of 2 groups (A or B) with 20 subjects each that received placebo or aspirin (100 mg/daily) for two weeks. At the end of the two week period (T15), patients of group A will be switched to placebo, while group B will be switched to aspirin for another 2 weeks (T30). Adherence will be confirmed by pill count at the end of each study period.
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Aspirin
- Aspirin (Active Comparator): Aspirin (100 mg/daily)
  Interventions: Drug: Aspirin

INTERVENTIONS:
Drug: Aspirin — Aspirin (100 mg once a day)

SUMMARY:
The specific research questions addressed in the present study are:

* to investigate the impact of treatment with low-dose aspirin in HIV-1-infected patients treated with ABC and test it would result in decreased in vivo platelet activation and platelet hyperreactivity
* to investigate if aspirin has the same effects in HIV-infected as in HIV-uninfected patients.

DETAILED DESCRIPTION:
Highly active antiretroviral therapy (HAART) may reduce the deleterious effects of HIV on the cardiovascular system by decreasing viral load and chronic inflammation; however some antiretrovirals enhance cardiovascular risk due to direct adverse effects on platelets or the endothelium.

Abacavir/lamivudine (ABC/3TC) and tenofovir/emtricitabine (TDF/FTC) are the most widely used nucleoside reverse transcriptase inhibitor (NRTI) associations in HAART. ABC has been initially considered as one of the most benign antiretroviral drugs due to a better metabolic profile than other nucleoside analogues, but since the D.A.D. study reported an association between the use of ABC and an increase in cardiovascular risk there has been controversy around this drug.

Clinical evidence suggests that in vivo platelet activation and platelet hyperreactivity contribute to adverse cardiovascular events and hyperreactive platelets may transform a normal reparative response to a mild arterial injury into an unwanted thrombotic event.

Aspirin is the cornerstone in the prevention of atherothrombotic events, as it has been shown to be effective both in the primary and secondary prevention of MI (6), and its beneficial effects likely involve the modulation of inflammatory and immune pathways. But despite heightened awareness regarding elevated CVD risk among HIV-infected patients, aspirin or others antiplatelet therapy were markedly underprescribed among HIV-infected patients at risk for CVD events (7).

Based on this, the proposed study will assess whether low-dose aspirin, in well-characterized HIV-1-infected patients treated with ABC, would result in decreased in vivo platelet activation and platelet hyperreactivity. Moreover will be investigate if aspirin will have the same effects in HIV-infected as in HIV-uninfected patients.

ELIGIBILITY:
Inclusion Criteria:

* a viral load <50 copies per millilitre
* ABC treatment for at least 6 months

Exclusion Criteria:

* age younger than 18
* nonsteroidal anti-inflammatory drug use in the past week (including aspirin), renal failure (creatinine clearance <30 mL/min), platelet count <100,000/microL, history of gastrointestinal bleeding within the last 6 months, presence of coexisting inflammatory disease, cancer, active bacterial or fungal infection, bleeding history, oral anticoagulant therapy and allergy to aspirin

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01-02 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-10-12 (Actual)

PRIMARY OUTCOMES:
Platelet reactivity | Change from baseline at day 15 and at day 30.
  PFA-100® collagen/epinephrine (C/EPI) cartridge closure time; light transmission aggregometry induced by arachidonic acid (1mM), collagen (0.8, 1.2 and 2 microg/ml) and epinephrine (100 microM); PAC-1; soluble P-selectin; sCD40L; platelet microparticles detection and quantification.

SECONDARY OUTCOMES:
Serum TxB2 levels and urinary 11-dehydro-TxB2 levels | Change from baseline at day 14 after aspirin intake.

IPD SHARING:
Plan to Share IPD: No